CLINICAL TRIAL: NCT01386008
Title: Evaluation of DW Silicone Hydrogel Lens Compared to DW Silicone Hydrogel Lens
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unexpected adverse events
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CV-10-50
Record Dates: First submitted 2011-05-22; First posted 2011-06-30 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- enfilcon A + senofilcon A (Other): Simultaneous wearing of daily wear contact lenses - investigational enfilcon A contact lenses in one eye and comparator senofilcon A worn in the other
  Interventions: Device: senfilcon A contact lens; Device: investigational enfilcon A

INTERVENTIONS:
Device: senfilcon A contact lens — senofilcon A spherical contact lens worn in a daily wear modality
Device: investigational enfilcon A — investigational enfilcon A, worn daily wear modality

SUMMARY:
The purpose of this study is to evaluate the performance of the investigational CooperVision silicone hydrogel lens compared to a currently-marketed silicone hydrogel contact lens up to 30 days of daily lens wear.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age as of the date of evaluation for the study.
2. Not using any ocular medications
3. Have a self-reported full eye examination within 2 years.
4. Have:

   * read the Informed Consent
   * be given an explanation of the Informed Consent
   * indicate understanding of the Informed Consent
   * signed the Informed Consent document.
5. Be willing and able to adhere to the instructions set forth in this protocol and able to keep all specified appointments.
6. Be an adapted, current full-time silicone hydrogel or soft contact lens wearer. An adapted full-time wearer is defined as wearing contact lenses on a daily basis for at least 8 hours per day for at least one month prior to participation in the study.
7. Possess wearable and visually functional eyeglasses.
8. Be in good general health, based on his/her knowledge.
9. Require spectacle lens powers between -1.00 and -6.00 diopters sphere with no more than 0.75 diopter of refractive astigmatism in order to have the best spherical equivalent power of -6.50 or less.
10. Be willing to wear contact lenses in both eyes.
11. Have manifest refraction Snellen visual acuities (VA) equal to or better than 20/25 (less than or equal to LogMAR 0.10) in each eye.
12. Upon completing the fitting process with the lenses to be worn in the study, have contact lens Snellen VA equal to or better than 20/30 in each eye.

Exclusion Criteria:

1. Wearing lenses in a monovision modality and is unwilling to be fit with distance lenses in both eyes. NOTE: Subjects may not wear lenses in a monovision modality at any time during the study as it will interfere with the visual acuity analysis.
2. Any active participation in another one-day clinical trial within 7 days prior to this study or another dispensing trial within 30 days prior to this study.
3. Currently pregnant (to the best of the subject's knowledge), is lactating or is planning a pregnancy within the next month.
4. Has a known sensitivity to ingredients used in the over the counter contact lens care approved for use in the study.
5. Previous refractive surgery/anterior segment surgery; or current or previous orthokeratology treatment or irregular cornea.
6. Is aphakic or pseudophakic.
7. Unable to achieve a satisfactory fit with the lens designs used in the study
8. Ocular or systemic disease such as, but not limited to: anterior uveitis or iritis (past or present), glaucoma, Sjögren's syndrome, lupus erythematosus, sclerodermia, keratoconus or type II diabetes.
9. The need for topical ocular medications or any medication which might contradict contact lens wear or which would require the lenses to be removed during the day.
10. The presence of clinically anterior segment infection, inflammations or abnormalities; such as iritis; or any infection of the eye, lids, or associated structures.
11. A history of herpetic keratitis.
12. A known history of corneal hypoesthesia (reduced corneal sensitivity) or active corneal ulcer, corneal infiltrates or fungal infection.
13. A history of papillary conjunctivitis that has interfered with contact lens wear.
14. Slit lamp findings that would contraindicate contact lens wear, including but not limited to:

    * Pathological dry eye or associated dry eye symptoms with decreased tear levels and punctuate staining > grade 2
    * Pterygium
    * Corneal scars within the visual axis
    * Corneal edema or corneal staining ≥ grade 2
    * Neovascularization or ghost vessels > 1.0 mm in from the limbus
    * Giant papillary conjunctivitis (GPC) of > grade 2.
    * Seborrheic eczema, seborrheic conjunctivitis or blepharitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Clinical Research Center, University of California, Berkeley, Berkeley, California, United States
- University of Manchester, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 28 recruited, 4 disqualified due to significant anterior ocular health findings, 4 passed screening and scheduled for lense fit/dispense when study discontinued.
Groups:
- Overall Study Group: Participants wear one enfilcon A (test) contact lens in one eye and one senofilcon A (comparator) contact lens in the other. Both lenses are worn daily wear.
Period: Overall Study
Arm/Group | Overall Study Group
Started | 20
Completed | 0
Not Completed | 20
Not completed — exited w/o incident /study discontinued | 17
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study Group
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4

OUTCOME MEASURES:

1. Secondary Outcome: Investigator Surface Preference
Description: Investigator Surface Preference rated on a linear scale (Lens assessment biomicroscopy: 1=strong R, 2=slight R, 3=No Pref, 4=slight L, 5=strong L)
Time Frame: V1 (Initial), V2 (Day-7), V3 (Day-14), V4 (Day-30)
Population: Not all subjects completed the study measures at each outcome measurement time frame before the study was terminated. 20 participants completed V1 and only 1 participant completed the V2 follow-up. V3 and V4 cannot be analyzed.
Measure: Number; unit: participants
Arm/Group | Enfilcon A + Senofilcon A
Number analyzed (Participants) | 20
participants
  Preferred Test Lens V1 | 6
  No Preference V1 | 5
  Preferred Control Lens V1 | 9
  Preferred Test Lens V2 | 0
  No Preference V2 | 1
  Preferred Control Lens V2 | 0

2. Primary Outcome: Subjective Comfort Preference - Participants Preference Response
Description: Subjective responses of participants administered by questionnaire and measured on a linear scale (0-100) measured at each visit.
Time Frame: V1 (Initial), V2 (Day-7), V3 (Day-14), V4 (Day-30)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Enfilcon A + Senofilcon A
Number analyzed (Participants) | 20
participants
  Preferred Test lens Visit 1 | 7
  No Preference Visit 1 | 8
  Preferred Control Lens Visit 1 | 5
  Preferred Test lens Visit 2 | 0
  No Preference Visit 2 | 1
  Preferred Control lens Visit 2 | 0

3. Primary Outcome: Ocular Health
Description: Ocular health determined by biomicroscopy recorded on a severity scale (0-4) for change from baseline over 30 days.
Time Frame: Change from baseline over 30 days measured at V1 (Initial), V2 (Day-7), V3 (Day-14), V4 (Day-30)
Population: Not all subjects completed the study measures at each outcome measurement time frame before the study was terminated. 20 participants completed V1 and only 1 participant completed the V2 follow-up. Change from baseline V1 over 30 days V4 cannot be analyzed.
Arm/Group | Enfilcon A + Senofilcon A
Number analyzed (Participants) | 0

4. Secondary Outcome: Investigator Fit Preference
Description: Investigator Fit Preference rated on a linear scale (Lens assessment biomicroscopy: 1=strong R, 2=slight R, 3=No Pref, 4=slight L, 5=strong L)
Time Frame: V1 (Initial), V2 (Day-7), V3 (Day-14), V4 (Day-30)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Enfilcon A + Senofilcon A
Number analyzed (Participants) | 20
participants
  Preferred Test Lens V1 | 7
  No Preference V1 | 10
  Preferred Control Lens V1 | 3
  Preferred Test Lens V2 | 1
  No Preference V2 | 0
  Preferred Control Lens V2 | 0

ADVERSE EVENTS:
Groups:
- Overall Study Group: investigational enfilcon A contact lenses worn daily wear and senofilcon A contact lens worn daily wear
Arm/Group | Overall Study Group
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study Group (N=20)
blurred vision (Eye disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Incomplete data sets / Data not analyzed / Not all subjects completed the study measures at each outcome measurement time frame before the study was terminated. 20 participants completed V1 and only 1 participant completed the V2 follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigators are not permitted to publish or make public any of the results without prior written approval from the Sponsor.